CLINICAL TRIAL: NCT07218731
Title: Presbyopic Wear Experience With Multifocal Lenses Compared to Single Vision Lenses and Reading Glasse
Brief Title: Presbyopic Wear Experience With Multifocal Lenses Compared to Single Vision Lenses and Reading Glasses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Fogt, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY20252007
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Presbyopia Correction; Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multifocal contact lenses (Active Comparator): multifocal contact lenses
  Interventions: Device: Multifocal contact lenses
- Spherical contact lenses with reading glasses (Active Comparator): spherical contact lenses used with reading glasses
  Interventions: Device: Spherical contact lenses

INTERVENTIONS:
Device: Multifocal contact lenses — Multifocal contact lenses
  Arms: Multifocal contact lenses
Device: Spherical contact lenses — spherical contact lenses
  Arms: Spherical contact lenses with reading glasses

SUMMARY:
The purpose of the study is to assess participant experience when wearing multifocal contact lenses compared to spherical contact lenses with reading glasses.

ELIGIBILITY:
Inclusion Criteria:

1. At least 40 years of age.
2. Ability to give informed consent.
3. Subjects must have corrected distance visual acuity in both eyes equivalent to 20/25 or better at the screening visit.
4. Require an add power of +0.75 D or greater when tested at 40cm.
5. Good general health defined by medication use that has not changed within the last 30 days and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the Investigator.

Exclusion Criteria:

1. Current or active inflammation or infection as determined by the Investigator.
2. Current eye disease, infection or inflammation that affects the surface of the eye such as but not limited to moderate or greater blepharitis and ocular allergy.
3. History of refractive surgery.
4. Known history of allergy or sensitivity to contact lens solutions and/or sodium fluorescein.
5. Is pregnant or lactating or planning a pregnancy during enrollment of the study.
6. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable.
7. Have been diagnosed with dry eye previously
8. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Preference Survey | 8 weeks
  Percentage of participants who prefer the multifocal lenses compared to spherical lenses with reading glasses.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared with other researchers.